CLINICAL TRIAL: NCT02448212
Title: A Phase 1 Receptor Occupancy Study Using Positron Emission Tomography to Investigate Novel Ligand [11C]TASP0410699 Alone and Following Single Oral Dose Administrations of TS-121 in Healthy Adult (Male) Subjects
Brief Title: Exploratory Study Using Positron Emission Tomography With TS-121 and [11C]TASP0410699 in Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical R&D Inc. (Industry)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TS121-US103
Record Dates: First submitted 2015-05-13; First posted 2015-05-19 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Healthy
Keywords: PET; Receptor Occupancy
MeSH Terms: interventions — TASP0410699; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PART 1 (Test/Retest) (Experimental): Dosing with [11C]TASP0410699 for PET imaging without dosing of TS-121
  Interventions: Drug: [11C]TASP0410699; Radiation: Positron Emission Tomography (PET)
- PART 2 (PET Receptor Occupancy Study) (Experimental): Dosing with [11C]TASP0410699 for PET imaging with dosing of TS-121
  Interventions: Drug: TS-121; Drug: [11C]TASP0410699; Radiation: Positron Emission Tomography (PET)

INTERVENTIONS:
Drug: TS-121 — Oral
  Arms: PART 2 (PET Receptor Occupancy Study)
Drug: [11C]TASP0410699 — Intravenous radiotracer
Radiation: Positron Emission Tomography (PET) — Imaging scanning procedure

SUMMARY:
The purpose of this study is to evaluate the binding of a novel tracer, [11C]TASP0410699, using Positron Emission Tomography (PET) scans with or without dosing of TS-121

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males 18 - 55 years of age (at time of initial informed consent)
2. Body weight ≥ 50 kg
3. Body Mass Index (BMI) 18 - 30 kg/m2
4. Male subjects with partners of childbearing potential must agree to use appropriate and effective measures of contraception for 90 days following drug administration

Exclusion Criteria:

1. Prescription, over-the-counter or herbal medications, supplements, within 14 days before the study.
2. Clinically significant abnormal electrocardiogram, physical examination, or hematology, biochemistry, hormone, or urinalysis values at screening & baseline.
3. Significant history &/or presence of hepatic, renal, cardiovascular, hemodynamic, pulmonary, gastrointestinal, hematological, CNS, immunologic, ophthalmologic, metabolic, endocrine, or oncological disease or condition within last 5 years.
4. Current use of tobacco or tobacco-containing products, recent history of alcohol or drug abuse OR positive urine screen for alcohol or controlled substances at screening or baseline.
5. History &/or current evidence of serologic positive results for hepatitis B or C, or HIV.
6. Donation or acute loss of 450 milliliters or more of blood or plasma, within 60 days of the study.
7. Any subject who has received treatment with a non-FDA approved drug within 30 days of study screening.
8. Subjects who suffer from claustrophobia.
9. Current, past, or anticipated exposure to radiation in the workplace or participation in other research studies involving ionizing radiation that would exceed the yearly dose limits for normal subjects.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Positron emission tomography measure (receptor occupancy) | Day 1 through Day 3

SECONDARY OUTCOMES:
Pharmacokinetic parameters of TS-121 | Day 1 through Day 3
  Area under the plasma concentration (AUC) from time zero to time of last measurable concentration
Pharmacokinetic parameters of TS-121 | Day 1 through Day 3
  Maximum concentration (Cmax)
Pharmacokinetic parameters of TS-121 | Day 1 through Day 3
  Time to attain cmax (Tmax)
Composite safety as assessed by clinical laboratory tests, 12-lead ECG, vital signs, adverse events and physical examinations | up to Day 11

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. Carson, Ph.D., Principal Investigator — Yale University; Shoji Yasuda, Study Director — Taisho Pharmaceutical R&D Inc.
Locations (1):
- Yale University PET Center, New Haven, Connecticut, United States